CLINICAL TRIAL: NCT03524794
Title: HepCare: The Effectiveness of Community Based Interventions With Peer Support to Improve Case Detection, Carry Out Pre-treatment Assessments and Assist Underserved Populations Through HCV Treatment
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: University College, London (Other)
Responsible Party: Sponsor
Other Study IDs: 17/0033
Record Dates: First submitted 2017-08-18; First posted 2018-05-15 (Actual); Last update posted 2018-05-18 (Actual); Status verified 2018-05

CONDITIONS: Hepatitis C; Infectious Disease
MeSH Terms: conditions — Hepatitis C; Communicable Diseases

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Hepatitis C infection is a major cause of chronic liver disease and death with approximately 3% of the world's population is infected with hepatitis C virus (HCV).

New drug therapies called new direct-acting antivirals (DAAs) have been developed and have proven to be well tolerated with minimal side effects. The current costs of these agents are extremely high, however, they provide an opportunity to cure most patients of HCV if they can access and adhere to treatment. The bigger challenge is to engage and cure underserved groups who are not accessing medical care, or who have other complex problems, including homelessness, incarceration, and substance misuse problems.

Strategies to improve HCV case detection and case management have much to learn from other infectious diseases. Tuberculosis (TB) disproportionately affects in large part the same group of individuals and community models of care have been used with great success. Strategies such as active case finding, community based screening and treatment, directly observed therapy (DOT) and peer support have all shown high rates of case detection and treatment completion.

These strategies are currently being used by the Find&Treat team, UCLH NHS Trust and this study will ain in evaluating it's effectiveness. Previously used to aid homeless patients engage with treatment services for TB, it is now being used with other disease groups such as HCV.

This observational study aims to assess the effectiveness of community based interventions with peer support to improve case detection, carry out pre-treatment assessments and assist underserved populations through HCV treatment by the Find&Treat service.

DETAILED DESCRIPTION:
1. Introduction

   Hepatitis C infection is a major cause of chronic liver disease and death throughout the world1. Approximately 3% of the world's population is infected with hepatitis C virus (HCV)2.

   HCV is transmitted by blood and in the UK occurs primarily through injecting drug use. Chronically infected people are at risk of progressive liver disease characterised by hepatocellular inflammation, hepatic fibrosis, cirrhosis and hepatocellular carcinoma (HCC). These complications develop only in a proportion of patients and only after many years or decades of infection3. It has been estimated that up to 20% of chronically infected individuals will develop cirrhosis of the liver over a 20 to 25 year period. Approximately 3% to 4% of patients with cirrhosis will develop HCC per year3.

   New drug therapies such as protease and polymerase inhibitors called direct-acting antivirals (DAAs) have been developed in the last ten years and have recently been licensed for use worldwide. These DAAs have proven to be very well tolerated with minimal, and sometimes no, side effects. The current costs of these agents are extremely high, limiting their use to select populations of infected patients. However, they provide an opportunity to cure most patients with HCV if they can access and adhere to treatment. A bigger challenge is to engage and cure those who are not accessing medical care, or who have other complex problems, including homelessness, incarceration, and substance misuse. These underserved populations are disproportionately affected by infectious diseases such as HCV and face many challenges to access testing and adherence to treatment.

   There has been previously demonstrated a high prevalence (13% RNA detectable HCV4) of chronic HCV infection among homeless people opportunistically screened at residential hostels and day centres across London. Data from the HALT Hepatitis Study5 showed that 41% of HCV Ab positive recruits were homeless at enrolment and that over 60% of HCV infected patients knew of their status but had disengaged from treatment services. This population therefore includes a high number of undiagnosed cases and previously known HCV positive cases who are not accessing treatment services.

   The epidemiology of HCV among homeless populations in the UK is poorly understood. Currently there are no data on the extent of liver fibrosis in this population to inform strategies for future management and estimate potential resource requirements to effectively mobilise treatment to this vulnerable and underserved group. Early detection of significant fibrosis is critical to prevent severe disease and death. Ongoing drug or alcohol use is not a contra-indication to hepatitis C treatment, and research shows that people who are actively using drugs can and should be treated for hepatitis C6. Point of care tests (POCTs) mean that infection can be identified immediately in the community reducing the risk of loss to follow up. Transient liver elastography (performed using FibroScan®) is now the gold standard in the assessment for liver fibrosis. FibroScanning is a 5 minute non-invasive, painless procedure to accurately assess liver fibrosis with high reproducibility7. This means that mush of what traditionally required several hospital appointments can now be done in potentially one outreach session.

   Strategies to improve HCV case detection and management have much to learn from the management of Tuberculosis (TB), a disease which affects the same group of individuals and community models of care have been used with great success. Strategies such as active case finding, community based screening and treatment, directly observed therapy (DOT) and peer support have all shown high rates of case detection and treatment completion.

   The Find&Treat Mobile Health Unit (MHU) from UCLH NHS Trust provides health screening for homeless individuals across various sites in London, UK such homeless hostels, day centres and drug services. They are experienced in using outreach models of care and peer advocates for infectious diseases such as TB to engage patients with specialist care. As HCV treatment moves into the community there is a need to evaluate outreach activities to inform future practice and care.
2. Aims and Objectives

   This study aims to assess the effectiveness of community based interventions with peer support to improve case detection, carry out pre-treatment assessments and assist underserved populations through HCV treatment by the Find&Treat service.

   Primary Objective

   Evaluate the effectiveness of the HCV community based detection and management including screening, liver assessment and treatment support in underserved populations using mobile health facilities and peer support.

   Secondary Objectives
   * Estimate the proportion of homeless people with chronic HCV infection and their degree of liver fibrosis.
   * Risk factors for HCV infection and for re-infection for those completing treatment or testing negative at recruitment.
   * Report this experience to inform the development of further programmes in the UK and other EU countries.
3. Study design

This is an observational study to establish the effectiveness of intensified community based screening, liver assessment and supported treatment for homeless people and underserved populations. Patients will be recruited from an NHS mobile health outreach service screening individuals accessing homeless and drug services in London, UK.

Following enrolment patient will be followed up for up to 12 months or until an appropriate defined clinical end point is reached. Successful engagement with community based HCV screening and treatment is defined as:

i. Successful pre-treatment assessment and a decision to not proceed by the clinician ii. Engagement with treatment support (including offered, start or completion of therapy according to individual circumstance)

Preliminary data from the HALT study (1) shows an effect size in improved engagement of 1.9. To detect a 20% increase in individuals successfully engaging with community services, from a baseline of 20%, we would need to recruit 164 individuals who are HCV positive (with 90% power and 5% significance level) compared with 82 in the comparison group. The clinical team would therefore have to screen 820 individuals assuming a rate of infection of 20%, which was found in previous pilot study work.

Among those screened we will calculate the prevalence of hepatitis C infection and the severity of disease in this population compared with published data and risk factors for chronic HCV infection and re-infection for those achieving SVR or test negative. We will also investigate the proportion completing treatment and factors associated with better treatment completion and SVR using multivariable regression models. Statistical software used in the analysis will be STATA version 14.1.

(1) The HALT Study. Unpublished: http://www.isrctn.com/ISRCTN24707359

ELIGIBILITY:
Inclusion Criteria:

* Over 16 years of age
* Underserved populations in the community. This is defined as groups whose social circumstances, language, culture or lifestyle make it difficult to access diagnostic and treatment services, self administer treatment or attend regular appointments for clinical follow up. This could include people who are homeless, people who misuse substances, prisoners, vulnerable migrants.
* Willingness and ability to provide signed informed consent
* The language ability to understand the PIS and other study information and therefore to able to provide informed consent

Exclusion Criteria:

* Less 16 years of age
* Unable to give informed consent

Min Age: 16 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: Underserved populations in the community. This is defined as groups whose social circumstances, language, culture or lifestyle make it difficult to access diagnostic and treatment services, self administer treatment or attend regular appointments for clinical follow up. This could include people who are homeless, people who misuse substances, prisoners, vulnerable migrants
Sampling Method: Non-Probability Sample
Enrollment: 164 (Estimated)
Dates: Start 2017-08-08 (Actual); Primary Completion 2018-12-31 (Estimated); Study Completion 2019-03-31 (Estimated)

PRIMARY OUTCOMES:
Successful engagement with community based HCV screening and treatment | 18 months
  Successful engagement with community based HCV screening and treatment is defined as:
  i. Successful pre-treatment assessment and a decision to not proceed by the clinician ii. Engagement with treatment support (including offered, start or completion of therapy according to individual circumstance)

SECONDARY OUTCOMES:
Estimate the proportion of homeless people with chronic HCV infection and their degree of liver fibrosis. | 18 months
  Estimate the proportion of homeless people with chronic HCV infection and their degree of liver fibrosis.
Risk factors for HCV infection and for re-infection for those completing treatment or testing negative at recruitment. | 18 months
  Risk factors for HCV infection and for re-infection for those completing treatment or testing negative at recruitment.

CONTACTS AND LOCATIONS:
Overall Officials: Alistair Story, Phd, Principal Investigator — University College London Hospital
Locations (1):
- University College London, London, United Kingdom

IPD SHARING:
Plan to Share IPD: No